CLINICAL TRIAL: NCT04512521
Title: FUNLUM: Functional Lung MRI for Early Treatment Response Assessment and Outcome Prediction for Patients With Severe Eosinophilic Asthma on Anti IL 5 Antibody Therapy
Brief Title: Functional Lung MRI for Early Treatment Response Assessment for Patients With Eosinophilic Asthma
Acronym: FUNLUM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 8832_BO_S_2020; 213598 (Other: GSK tracking number)
Record Dates: First submitted 2020-07-29; First posted 2020-08-13 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Asthma; Eosinophilic
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood eosinophil cell count, IgE FENO capillary BGA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- eosinophilic asthma
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab therapy

SUMMARY:
Patients with severe eosinophilic asthma will be placed on biologics if they continue to be uncontrolled despite maximized inhalation therapy or if they are only controlled under oral corticosteroids. Among biologics, 80% of patients respond to treatment and improve clinically, but approximately 20% are non-responders and up to date no established predictive factors for treatment response exist. Among the responders, about 30% respond very well (so-called super responders), the rest shows moderate improvements. As the lung function, one main criterion to evaluate treatment response improves in most patients with delay, the response (or non-response) to treatment can only be reliably estimated after 4 to 12 months. This can lead to prolonged use of medication in non-responders (overtreatment) on one hand and to unjustified and premature termination of therapy (undertreatment) on the other hand (GINA report 2019).

Functional lung MRI has the potential to show early changes in lung microstructure, regional ventilation and perfusion and thus has the potential for early detection of therapy response. Very promising results of dynamic regional ventilation and perfusion mapping using phase resolved functional lung (PREFUL) MRI have been shown recently.

However, if functional lung MRI can reliably detect treatment effects under Mepolizumab therapy and can help to predict a long-term patient outcome is still unknown. As these findings could directly influence clinical decision making this question is of high clinical relevance.

DETAILED DESCRIPTION:
Asthma is a chronic disease and affects approximately 300 million people worldwide. Of these patients 3-10% have severe asthma which is defined as asthma remaining uncontrolled despite treatment with high-dose inhaled glucocorticoids combined with other controllers (long-acting β2-agonist, long-acting antimuscarinic agent, leukotriene receptor antagonist or theophylline) and/or treatment with systemic glucocorticoids for at least 6 months. Severe asthma causes a high amount of medical expenses in asthma. For patients suffering from severe uncontrolled asthma, an IL-5 antibody (mepolizumab) has been approved for therapy when a type 2 inflammation was present. Treatment is well tolerated and a significant reduction of exacerbations, oral glucocorticoid use was reported. Another IL-5 antibody (reslizumab) and an IL-5 receptor antibody (benralizumab) are available now.

Patients with severe eosinophilic asthma will be placed on biologics if they continue to be uncontrolled under maximal therapy or if they are only controlled under oral corticosteroids. Among biologics, 80% of patients improve, 20% are non-responders, but there is no way to identify them early. Among the responders, about 30% respond very well (so-called super responders), the rest shows moderate improvements. The main problems at the moment are that lung function improvements are only delayed, the response (or non-response) can only be reliably estimated after 4 to 12 months. This leads on the one hand to prolonged use of medication in non-responders (overtreatment), on the other hand to unjustified and premature termination of therapy (undertreatment) (GINA report 2019).

Study Rationale Functional lung MRI has the potential to show early changes in lung microstructure, regional ventilation and perfusion and thus has the potential for early detection of therapy response. Very promising results of dynamic regional ventilation and perfusion mapping using phase resolved functional lung (PREFUL) MRI have been shown recently. This technique holds the promise to mature into a patient friendly sensitive MRI spirometry test, with novel clinically relevant information to guide clinical decision making and improve patient monitoring. PREFUL MRI typically uses standard 1.5T or 3T MRI equipment and is based on a routine gradient echo fast low angle shot (FLASH) sequence. PREFUL is well suited also for children, because it is a free breathing exam without the need for i.v. contrast and has a relatively short examination time. The ventilation, perfusion and dynamic flow-volume loop maps are reconstructed entirely after the image acquisition using complex registration and post processing algorithms developed and validated at Hannover Medical School. Preliminary unpublished data show that PREFUL MRI may detect changes in regional ventilation 3 months after anti IL 5 antibody therapy treatment.

However, if functional lung MRI can reliably detect changes at 3 months of Mepolizumab treatment and can predict long term patient outcome is still unknown, which is of high clinical relevance for future clinical decision making.

The aim of this study is to examine if early treatment changes of Mepolizumab treatment can be detected at 3 months measured by functional lung MRI and predict clinical outcome at 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent.
* Male and female subjects, aged ≥ 18 years.
* Patients which are eligible for treatment using anti-IL-5 -antibody treatment following guidelines: severe eosinophilic asthma and blood eosinophils of ≥150 cells/μL at screening or ≥ 300 cells/μL within 12 months prior to treatment
* Physician-diagnosed severe asthma according to ERS/ATS guidelines
* Treatment with a total daily dose of medium or high-dose ICS (e.g. ≥ 500μg fluticasone propionate, ≥ 800μg budesonide or equivalent total daily dose). ICS can be contained within an ICS/LABA combination product.
* At least one additional maintenance asthma controller e.g. LABA, LTRA, theophylline, LAMA, etc. with or without OCS

Exclusion Criteria:

* Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis, vital signs, lung function at screening visit, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study, or the subject's ability to participate in the study.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease other than Asthma (including but not confined to tuberculosis, bronchiectasis, cystic fibrosis, pulmonary hypertension, sarcoidosis, interstitial lung disease or lung fibrosis).
* History of drug or alcohol abuse.
* Risk of non-compliance with study procedures.
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
* History of an acute respiratory infection four weeks prior to enrolment. These patients will not be eligible, but will be permitted to be rescreened 4 weeks after the resolution of the respiratory tract infection.
* Subjects with severe renal impairment (GFR ≤ 30 mL/min) including those with end-stage renal disease requiring dialysis or urinary retention.
* Subjects with active/ clinical history of COPD.
* Subjects unable to undergo MRI scans, including claustrophobia or presence of any metal objects within the patient, preventing from MRI scan (e.g. pacemaker, aneurysm clips).
* History of asthma exacerbation that required treatment with antibiotics, systemic steroids (oral or intravenous) or hospitalization within 3 months prior to enrolment.
* Subjects with a body mass index (BMI) of more than 35 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be selected for this study consecutively by Dr. Suhling (or colleagues; Dr. Drick) from his Asthma outpatient clinic according to his clinical judgement.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-05-04 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Baseline ventilation-defect percentage by pulmonary MRI | baseline
  Baseline airway function by measuring ventilation-defect percentage by pulmonary MRI.
Ventilation-defect percentage by pulmonary MRI after 3 months treatment with Mepolizumab | 3 months
  To study the effect of Mepolizumab treatment after 3 months treatment compared to baseline on airway function by measuring ventilation-defect percentage by pulmonary MRI.
Baseline perfusion-defect percentage by pulmonary MRI | baseline
  Baseline vascular function by measuring pulmonary perfusion-defect percentage by pulmonary MRI
Perfusion-defect percentage by pulmonary MRI after 3 months treatment with Mepolizumab | 3 months
  To study the effect of Mepolizumab treatment after 3 months treatment compared to baseline on vascular function by measuring pulmonary perfusion-defect percentage by pulmonary MRI
Baseline ventilation/Perfusion mismatch by pulmonary MRI | baseline
  Baseline Ventilation/Perfusion match and mismatch measured by pulmonary MRI.
Ventilation/Perfusion mismatch by pulmonary MRI after 3 months treatment with Mepolizumab | 3 months
  To study the effect of Mepolizumab treatment after 3 months treatment compared to baseline as Ventilation/Perfusion match and mismatch measured by pulmonary MRI.

SECONDARY OUTCOMES:
Ventilation-defect percentage by pulmonary MRI after 6 weeks treatment with Mepolizumab | 6 weeks
  To study the effect of Mepolizumab treatment after 6 weeks treatment compared to baseline on airway function by measuring ventilation-defect percentage by pulmonary MRI.
Perfusion-defect percentage by pulmonary MRI after 6 weeks treatment with Mepolizumab | 6 weeks
  To study the effect of Mepolizumab treatment after 6 weeks treatment compared to baseline on airway function by measuring perfusion-defect percentage by pulmonary MRI.
Ventilation/Perfusion mismatch by pulmonary MRI after 6 weeks treatment with Mepolizumab | 6 weeks
  To study the effect of Mepolizumab treatment after 6 weeks treatment compared to baseline on airway function by measuring ventilation/perfusion mismatch by pulmonary MRI.
Baseline asthma control test | baseline
  Baseline airway function measured by asthma control test (ACT)
Asthma control test after 12 months of treatment with Mepolizumab | 12 months
  To study the effect of Mepolizumab treatment after 12 months compared to baseline on airway function measured by asthma control test (ACT).
Baseline Clinical lung function | baseline
  Baseline airway function measured by Clinical lung function via bodyplesmography
Clinical lung function after 12 months of treatment with Mepolizumab | 12 months
  To study the effect of Mepolizumab treatment after 12 months compared to baseline on airway function measured by Clinical lung function via bodyplesmography
Baseline fractional exhaled nitric oxide | baseline
  Baseline airway function measured by fractional exhaled nitrix oxide (FeNO)
Fractional exhaled nitric oxide after 12 months of treatment with Mepolizumab | 12 months
  To study the effect of Mepolizumab treatment after 12 months compared to baseline on airway function measured by fractional exhaled nitrix oxide (FeNO)
Baseline capillary blood gas analysis | baseline
  Baseline airway function measured by capillary blood gas analysis
Capillary blood gas analysis after 12 months of treatment with Mepolizumab | 12 months
  To study the effect of Mepolizumab treatment after 12 months compared to baseline on airway function measured by capillary blood gas analysis
Baseline blood eosinophil cell count | baseline
  Baseline airway function measured by blood eosinophil cell count
Blood eosinophil cell count after 12 months of treatment with Mepolizumab | 12 months
  To study the effect of Mepolizumab treatment after 12 months compared to baseline on airway function measured by blood eosinophil cell count
Baseline exacerbation rate | baseline
  Baseline airway function measured by exacerbation rate
Exacerbation rate after 12 months of treatment with Mepolizumab | 12 months
  To study the effect of Mepolizumab treatment after 12 months compared to baseline on airway function measured by exacerbation rate

CONTACTS AND LOCATIONS:
Overall Officials: Jens Vogel-Claussen, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] To T, Stanojevic S, Moores G, Gershon AS, Bateman ED, Cruz AA, Boulet LP. Global asthma prevalence in adults: findings from the cross-sectional world health survey. BMC Public Health. 2012 Mar 19;12:204. doi: 10.1186/1471-2458-12-204. PMID 22429515
- [Background] Hekking PW, Wener RR, Amelink M, Zwinderman AH, Bouvy ML, Bel EH. The prevalence of severe refractory asthma. J Allergy Clin Immunol. 2015 Apr;135(4):896-902. doi: 10.1016/j.jaci.2014.08.042. Epub 2014 Oct 16. PMID 25441637
- [Background] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Background] Braman SS. The global burden of asthma. Chest. 2006 Jul;130(1 Suppl):4S-12S. doi: 10.1378/chest.130.1_suppl.4S. PMID 16840363
- [Background] Pavord ID, Korn S, Howarth P, Bleecker ER, Buhl R, Keene ON, Ortega H, Chanez P. Mepolizumab for severe eosinophilic asthma (DREAM): a multicentre, double-blind, placebo-controlled trial. Lancet. 2012 Aug 18;380(9842):651-9. doi: 10.1016/S0140-6736(12)60988-X. PMID 22901886
- [Background] Mepolizumab treatment in patients with severe eosinophilic asthma. N Engl J Med. 2015 Apr 30;372(18):1777. doi: 10.1056/NEJMx150017. Epub 2015 Apr 10. No abstract available. PMID 25860645
- [Background] Bel EH, Wenzel SE, Thompson PJ, Prazma CM, Keene ON, Yancey SW, Ortega HG, Pavord ID; SIRIUS Investigators. Oral glucocorticoid-sparing effect of mepolizumab in eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1189-97. doi: 10.1056/NEJMoa1403291. Epub 2014 Sep 8. PMID 25199060
- [Background] Castro M, Zangrilli J, Wechsler ME, Bateman ED, Brusselle GG, Bardin P, Murphy K, Maspero JF, O'Brien C, Korn S. Reslizumab for inadequately controlled asthma with elevated blood eosinophil counts: results from two multicentre, parallel, double-blind, randomised, placebo-controlled, phase 3 trials. Lancet Respir Med. 2015 May;3(5):355-66. doi: 10.1016/S2213-2600(15)00042-9. Epub 2015 Feb 23. PMID 25736990
- [Background] Nair P, Wenzel S, Rabe KF, Bourdin A, Lugogo NL, Kuna P, Barker P, Sproule S, Ponnarambil S, Goldman M; ZONDA Trial Investigators. Oral Glucocorticoid-Sparing Effect of Benralizumab in Severe Asthma. N Engl J Med. 2017 Jun 22;376(25):2448-2458. doi: 10.1056/NEJMoa1703501. Epub 2017 May 22. PMID 28530840
- [Background] Voskrebenzev A, Gutberlet M, Klimes F, Kaireit TF, Schonfeld C, Rotarmel A, Wacker F, Vogel-Claussen J. Feasibility of quantitative regional ventilation and perfusion mapping with phase-resolved functional lung (PREFUL) MRI in healthy volunteers and COPD, CTEPH, and CF patients. Magn Reson Med. 2018 Apr;79(4):2306-2314. doi: 10.1002/mrm.26893. Epub 2017 Aug 30. PMID 28856715
- [Background] Kaireit TF, Gutberlet M, Voskrebenzev A, Freise J, Welte T, Hohlfeld JM, Wacker F, Vogel-Claussen J. Comparison of quantitative regional ventilation-weighted fourier decomposition MRI with dynamic fluorinated gas washout MRI and lung function testing in COPD patients. J Magn Reson Imaging. 2018 Jun;47(6):1534-1541. doi: 10.1002/jmri.25902. Epub 2017 Nov 21. PMID 29160020
- [Background] Kaireit TF, Voskrebenzev A, Gutberlet M, Freise J, Jobst B, Kauczor HU, Welte T, Wacker F, Vogel-Claussen J. Comparison of quantitative regional perfusion-weighted phase resolved functional lung (PREFUL) MRI with dynamic gadolinium-enhanced regional pulmonary perfusion MRI in COPD patients. J Magn Reson Imaging. 2019 Apr;49(4):1122-1132. doi: 10.1002/jmri.26342. Epub 2018 Oct 22. PMID 30350440
- [Background] Klimes F, Voskrebenzev A, Gutberlet M, Kern A, Behrendt L, Kaireit TF, Czerner C, Renne J, Wacker F, Vogel-Claussen J. Free-breathing quantification of regional ventilation derived by phase-resolved functional lung (PREFUL) MRI. NMR Biomed. 2019 Jun;32(6):e4088. doi: 10.1002/nbm.4088. Epub 2019 Mar 25. PMID 30908743
- [Background] Bauman G, Puderbach M, Deimling M, Jellus V, Chefd'hotel C, Dinkel J, Hintze C, Kauczor HU, Schad LR. Non-contrast-enhanced perfusion and ventilation assessment of the human lung by means of fourier decomposition in proton MRI. Magn Reson Med. 2009 Sep;62(3):656-64. doi: 10.1002/mrm.22031. PMID 19585597
- [Background] Moher Alsady T, Voskrebenzev A, Greer M, Becker L, Kaireit TF, Welte T, Wacker F, Gottlieb J, Vogel-Claussen J. MRI-derived regional flow-volume loop parameters detect early-stage chronic lung allograft dysfunction. J Magn Reson Imaging. 2019 Dec;50(6):1873-1882. doi: 10.1002/jmri.26799. Epub 2019 May 27. PMID 31134705
- [Background] Svenningsen S, Eddy RL, Lim HF, Cox PG, Nair P, Parraga G. Sputum Eosinophilia and Magnetic Resonance Imaging Ventilation Heterogeneity in Severe Asthma. Am J Respir Crit Care Med. 2018 Apr 1;197(7):876-884. doi: 10.1164/rccm.201709-1948OC. PMID 29313707
- [Background] Gutberlet M, Kaireit TF, Voskrebenzev A, Lasch F, Freise J, Welte T, Wacker F, Hohlfeld JM, Vogel-Claussen J. Free-breathing Dynamic 19F Gas MR Imaging for Mapping of Regional Lung Ventilation in Patients with COPD. Radiology. 2018 Mar;286(3):1040-1051. doi: 10.1148/radiol.2017170591. Epub 2017 Oct 3. PMID 28972817
- [Background] Couch MJ, Ball IK, Li T, Fox MS, Biman B, Albert MS. 19 F MRI of the Lungs Using Inert Fluorinated Gases: Challenges and New Developments. J Magn Reson Imaging. 2019 Feb;49(2):343-354. doi: 10.1002/jmri.26292. Epub 2018 Sep 24. PMID 30248212
- [Background] Horn FC, Marshall H, Collier GJ, Kay R, Siddiqui S, Brightling CE, Parra-Robles J, Wild JM. Regional Ventilation Changes in the Lung: Treatment Response Mapping by Using Hyperpolarized Gas MR Imaging as a Quantitative Biomarker. Radiology. 2017 Sep;284(3):854-861. doi: 10.1148/radiol.2017160532. Epub 2017 May 4. PMID 28471738
- [Background] Capaldi DPI, Sheikh K, Eddy RL, Guo F, Svenningsen S, Nair P, McCormack DG, Parraga G; Canadian Respiratory Research Network. Free-breathing Functional Pulmonary MRI: Response to Bronchodilator and Bronchoprovocation in Severe Asthma. Acad Radiol. 2017 Oct;24(10):1268-1276. doi: 10.1016/j.acra.2017.04.012. Epub 2017 May 24. PMID 28551402
- [Background] Svenningsen S, Kirby M, Starr D, Leary D, Wheatley A, Maksym GN, McCormack DG, Parraga G. Hyperpolarized (3) He and (129) Xe MRI: differences in asthma before bronchodilation. J Magn Reson Imaging. 2013 Dec;38(6):1521-30. doi: 10.1002/jmri.24111. Epub 2013 Apr 15. PMID 23589465
- [Background] Vogel-Claussen J, Schonfeld CO, Kaireit TF, Voskrebenzev A, Czerner CP, Renne J, Tillmann HC, Berschneider K, Hiltl S, Bauersachs J, Welte T, Hohlfeld JM. Effect of Indacaterol/Glycopyrronium on Pulmonary Perfusion and Ventilation in Hyperinflated Patients with Chronic Obstructive Pulmonary Disease (CLAIM). A Double-Blind, Randomized, Crossover Trial. Am J Respir Crit Care Med. 2019 May 1;199(9):1086-1096. doi: 10.1164/rccm.201805-0995OC. PMID 30641027
- [Background] Hueper K, Parikh MA, Prince MR, Schoenfeld C, Liu C, Bluemke DA, Dashnaw SM, Goldstein TA, Hoffman EA, Lima JA, Skrok J, Zheng J, Barr RG, Vogel-Claussen J. Quantitative and semiquantitative measures of regional pulmonary microvascular perfusion by magnetic resonance imaging and their relationships to global lung perfusion and lung diffusing capacity: the multiethnic study of atherosclerosis chronic obstructive pulmonary disease study. Invest Radiol. 2013 Apr;48(4):223-30. doi: 10.1097/RLI.0b013e318281057d. PMID 23385398
- [Background] Eddy RL, Svenningsen S, McCormack DG, Parraga G. What is the minimal clinically important difference for helium-3 magnetic resonance imaging ventilation defects? Eur Respir J. 2018 Jun 28;51(6):1800324. doi: 10.1183/13993003.00324-2018. Print 2018 Jun. No abstract available. PMID 29650564
- [Background] Drick N, Seeliger B, Welte T, Fuge J, Suhling H. Anti-IL-5 therapy in patients with severe eosinophilic asthma - clinical efficacy and possible criteria for treatment response. BMC Pulm Med. 2018 Jul 18;18(1):119. doi: 10.1186/s12890-018-0689-2. PMID 30021546